CLINICAL TRIAL: NCT05026515
Title: The Influence of Parental Behavior on the Course of the Pediatric Dentistry : a Prospective Study
Brief Title: The Influence of Parental Behavior on the Course of the Pediatric Dentistry Session
Status: Completed | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Tania Vanhée, Pediatric Dentist, Université Libre de Bruxelles
Other Study IDs: O.M. 007
Record Dates: First submitted 2021-04-24; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Behavior, Child; Parents; Dental Anxiety
MeSH Terms: conditions — Child Behavior | interventions — Single Parent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 4 years and under: Children coming at dental appointment, aged 4 years and under
  Interventions: Behavioral: Parents
- 5 to 6 years: Children coming at dental appointment, aged 5 to 6 years
  Interventions: Behavioral: Parents
- 7 years and over: Children coming at dental appointment, aged 7 years and over
  Interventions: Behavioral: Parents

INTERVENTIONS:
Behavioral: Parents — To observe the influence of the parents/caregivers behavior on their child during dental treatment

SUMMARY:
The aim of the experiment is to analyze the impact of the behavior of the accompanying parent on the behavior of the child during a first dental session according to the age group.

DETAILED DESCRIPTION:
I will receive the children for consultation at the CHU Saint Pierre - César de Paepe site, to assess the impact of parents' behavior on the child.

First, I will make a first contact with the child in the waiting room using the CORAH scale (self-assessment based on diagrams) which will allow him to assess his temperament in the face of dental care. . Then, I will have the parents / caregiver sign informed consent and authorization to film.

Once the child enters the practice, the video recording will be initiated: the installation on the seat, the confidence building and the care provided will be filmed.

These videos will then be analyzed by several practitioners from different categories (experts in pedodontics, general dentists, dental students, etc.) using the Venham hetero-assessment scale modified for the behavior of the child and of a scale of parental cooperation. These practitioners will be selected via the ADUB (association of dentists of Université Libre de Bruxelles) and some of them could be external to the hospital.

Following this study, the results obtained will be described and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* be in the correct age group and agree to participate in the study

Exclusion Criteria:

* not be in the right age group, refuse to participate in the study

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 60 patients presenting for the first time to the pediatric dentistry consultation at the CHU Saint-Pierre - César de Paepe site were selected for this study between. 3 groups of 20 children, respectively aged 4 and under, 5 to 6 years old and over 7 years old, were formed.67 children participated in this study. They were divided into 3 groups according to their age (4 years and under, 5 to 6 years and 7 years and over). During the search, 7 patients were excluded: due to the image rights not granted. The data were collected and analyzed by 2 observers. Then a randomization took place thus creating a sample of 15 children divided into 3 same groups. The data were collected and analyzed by 20 practitioner observers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Parent behavior/Child Behavior | Two weeks
  By hetero-evaluation scale, 20 dentists will estimate the behavior of parents and children. The measurements via the observation of filmed sessions were carried out thanks to two views.

CONTACTS AND LOCATIONS:
Overall Officials: Tania Vanhee, DDS, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Tania Vanhée, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No